CLINICAL TRIAL: NCT02168764
Title: Sphenopalatine Ganglion Stimulation for the Treatment of Chronic Cluster Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Autonomic Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pathway CH-2
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Both arms of the study receive the ATI Neurostimulation System. Subjects are implanted with the ATI Neurostimulator and instructed to use the ATI Remote Controller to treat cluster attacks of at least moderate intensity by stimulating for 15 minutes before using any acute medications.
  Interventions: Device: ATI Neurostimulation System
- Control (Active Comparator): Both arms of the study receive the ATI Neurostimulation System. Subjects are implanted with the ATI Neurostimulator and instructed to use the ATI Remote Controller to treat cluster attacks of at least moderate intensity by stimulating for 15 minutes before using any acute medications.
  Interventions: Device: ATI Neurostimulation System

INTERVENTIONS:
Device: ATI Neurostimulation System — All subjects will be implanted with the ATI Neurostimulator which, along with the ATI Remote Controller, provides electrical stimulation.

SUMMARY:
The primary objective of the study is to demonstrate the safety and efficacy of SPG stimulation with the ATI Neurostimulation System when used to treat acute cluster attacks in chronic cluster headache patients.

ELIGIBILITY:
Inclusion Criteria:

* Age from ≥22 years old.
* Subject has been diagnosed with chronic cluster headache according to the 2013 ICHD, 3rd edition (beta version), criterion 3.1.2.
* Subject reports a minimum of 4 cluster attacks per week on the side of their dominant headache laterality. Subjects who report more than 8 attacks per day or attack duration of less than 30 minutes (untreated or unsuccessfully treated) must have been tested to rule out other forms of trigeminal autonomic cephalalgias.
* Both subject and physician judge previously or currently used preventive and/or acute cluster headache treatment to be inadequate.
* Subject is able to distinguish cluster attacks from other headaches (i.e., migraine, tension-type headaches).
* Subject agrees to not use therapy involving TENS or magnetic field treatment while the Neurostimulator is implanted.
* Subject agrees to not participate in supplemental or alternative therapy, including acupuncture and spinal manipulation, from Study Enrollment through the end of the Experimental Period of the study.
* Subject agrees to maintain current preventive headache medication regimens (no change in type, frequency, or dose) - except to manage tolerability - from Study Enrollment through the Experimental Period of the study.
* Subject agrees not to use any acute medications, including oxygen therapy, for their treatable cluster attacks during the Experimental Period until after they have used SPG stimulation therapy for at least 15 minutes.
* Subject has had a dental examination and cleaning in the past six (6) months.
* Subject has the ability to read and comprehend, and to reliably record information as required by the Protocol.
* Subject is able to provide written informed consent prior to participation in the study.

Exclusion Criteria:

* Subject's overall health, age and/or comorbidities place subject at high risk for complications from surgery and/or general anesthesia.
* Subject has had a change in type, dosage or dose frequency of preventive headache medications < one (1) month prior to study enrollment
* Subject has been diagnosed with any other form of Trigeminal Autonomic Cephalalgias (e.g., paroxysmal hemicrania, SUNCT, etc.) or has a history of trigeminal neuralgia.
* Subject has undergone facial surgery in the area of the pterygopalatine fossa or zygomaticomaxillary buttress ipsilateral to the planned implant site that, in the opinion of the Investigator, may lead to an inability to properly implant the Neurostimulator.
* Subject currently has an active oral or dental abscess or an active maxillary sinus infection based on present symptoms.
* Subject has been treated with therapeutic radiation to the facial region.
* Subject has been diagnosed with any major infectious processes such as osteomyelitis, or primary or secondary malignancies involving the face that have been active or required treatment in the past six (6) months.
* Subject has other significant pain problem(s) that, in the opinion of the Investigator, might confound the study assessments.
* Subject is a woman of childbearing potential who is pregnant, nursing, or not using contraception.
* Subject is currently participating or has participated in the last month in another clinical study in which the subject has, is, or will be exposed to an investigational or non-investigational drug or device.
* Subject has demonstrated or is believed to be at risk of non-compliance with study procedures (e.g., for completing the diary or maintaining a stable headache medicine regimen or returning for required follow-up visits).
* Subject is at risk of being unable to complete at least 1 year of follow-up (e.g., has plans to relocate).
* Subject has had previous lesional radio-frequency (RF) ablation, balloon compression, gamma knife, or glycerol treatments of the ipsilateral sphenopalatine ganglion (SPG), trigeminal ganglion or any branch of the trigeminal nerve.
* Subject has had blocks or non-lesional pulsed RF of the ipsilateral SPG in the last three (3) months.
* Subject's pterygomaxillary fissure is less than 1.2 mm in width at the level of the vidian canal, as determined by CT scan.
* Subject has undergone onabotulinumtoxinA injections of the head and/or neck or has had an occipital nerve block in the last three (3) months.
* Subject has or requires an active implanted medical device, such as a pacemaker/defibrillator, other neurostimulator, or cochlear implant.
* Subject is expected to require diathermy, electroconvulsive therapy (ECT), or transcranial magnetic stimulation (TMS).
* Subject has a history of bleeding disorders or coagulopathy and is unable to discontinue anticoagulation, antiplatelet, or GP IIb IIIa inhibitor medication in preparation for the implantation procedure.
* In the opinion of the Investigator, the subject currently meets criteria as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) for an active major depressive episode or for active significant psychiatric disorders, including dementia, uncontrolled general anxiety disorder, psychotic disorders or uncontrolled bipolar disorder. Exclusion criteria also include: active psychosis, untreated severe anxiety disorder, homicidal ideation, significant Axis II disorders and significant untreated sleep disorders.
* Subject currently has clinically significant drug or alcohol abuse as defined by DSM-IV-TR or is unable to refrain from substance abuse throughout the study.
* Subject has a history of malignancy or any other condition that requires MRI monitoring.
* Subject has a history of allergic or hypersensitive reactions to titanium, platinum, or implant grade silicone-polyurethane copolymers.
* Subject may be, in the opinion of the Investigator, at greater risk of infection (e.g., subjects with diabetes, taking steroids, with gingivitis/periodontitis, malnutrition or anorexia/bulimia) or at higher risk of harm from infections.
* Subject is currently using a tobacco cessation regimen (e.g. Wellbutrin, Zyban, Aplenzin, etc.).
* Subject is not suitable for the study for any reason (including overall health, pre-existing conditions or medications) in the judgment of the Investigator.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-07; Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Primary Safety | One year post-implant
  Characterization of all serious adverse events in all subjects who undergo an implantation procedure, through the completion of the Open Label Period.
Primary Efficacy | 28 weeks post-implant
  Compared between the two study arms: Proportion of stimulation-treated ipsilateral cluster attacks that achieve pain relief at 15 minutes following the start of stimulation without the use of acute medications prior to that time point.

SECONDARY OUTCOMES:
Secondary Efficacy | 28 weeks post-implant
  Compared between the two study arms: Proportion of stimulation-treated ipsilateral cluster attacks that achieve pain freedom at 15 minutes following the start of stimulation without the use of acute medications prior to that time point.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Goadsby, MD, PhD, Principal Investigator — UCSF Medical Center, Headache Center; David W Dodick, MD, Principal Investigator — Mayo Clinic, Department of Neurology
Locations (24):
- United States (24):
  - Mayo Clinic, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Stanford University, Stanford, California
  - Yale University, New Haven, Connecticut
  - New England Institute for Clinical Research, Stamford, Connecticut
  - University of Chicago, Illinois - SURGICAL CENTER ONLY, NOT AN ENROLLING CENTER, Chicago, Illinois
  - Diamond Headache Clinic, Chicago, Illinois
  - Robbins Headache Clinic, Northbrook, Illinois
  - Norton Neurology Services, Louisville, Kentucky
  - New England Regional Headache Center, Worcester, Massachusetts
  - Michigan Headache and Neurological Institute, Ann Arbor, Michigan
  - Headache Care Center (Springfield), Springfield, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Nevada Headache Institute, Las Vegas, Nevada
  - Dartmouth Hitchcock-Medical Center, Lebanon, New Hampshire
  - Dent Neurosciences Research Institute, Amherst, New York
  - Lenox Hill Hospital, The New York Head and Neck Institute - SURGICAL CENTER ONLY, NOT AN ENROLLING CENTER, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Island Neurological Association, Plainview, New York
  - Carolina Headache Institute, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Jefferson Headache Center, Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Texas, Southwestern, Dallas, Texas
  - Inova Medical Group Neurology and Headache, Falls Church, Virginia

REFERENCES:
- [Derived] Goadsby PJ, Sahai-Srivastava S, Kezirian EJ, Calhoun AH, Matthews DC, McAllister PJ, Costantino PD, Friedman DI, Zuniga JR, Mechtler LL, Popat SR, Rezai AR, Dodick DW. Safety and efficacy of sphenopalatine ganglion stimulation for chronic cluster headache: a double-blind, randomised controlled trial. Lancet Neurol. 2019 Dec;18(12):1081-1090. doi: 10.1016/S1474-4422(19)30322-9. PMID 31701891